CLINICAL TRIAL: NCT00732628
Title: Technical and Clinical Outcomes Following Placement of Boomerang Percutaneous Closure Device After Cerebral Angiography or Neurointerventional Procedures
Brief Title: Evaluating Outcomes in the Placement of Boomerang Percutaneous Device
Status: Terminated | Type: Observational
Why Stopped: Physician is no longer associated with the Univ. of Michigan Medical Center
Sponsor: University of Michigan (Other)
Responsible Party: Sameer Ansari MD, University of Michigan
Other Study IDs: HUM13883
Record Dates: First submitted 2008-07-25; First posted 2008-08-12 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Medical Device; Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Boomerang percutaneous closure unit: patients having a Boomerang percutaneous closure device after a Neurointerventional study
  Interventions: Device: Boomerang closure device

INTERVENTIONS:
Device: Boomerang closure device — Use of percutaneous of Boomerang closure device. Follow up outcomes evaluated after the use of Boomerang closure device.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Boomerang percutaneous closure device following diagnostic cerebral angiography or neurointerventional procedures.

Background:

Very few publications have evaluated this relatively novel percutaneous closure device.

DETAILED DESCRIPTION:
The purpose of this study is to document our experiences using the Boomerang closure device. Several different closure devices are used in the department of Radiology. A closure device is something that is placed in the artery in the leg just prior to removing the catheters from your leg at the end of the imaging or treatment procedure that is to be performed in the Department of Radiology. The devices used are all FDA approved. This study will compare the Boomerang device (a newer FDA approved device) to the other older devices currently being used. You may not have the Boomerang device used in your procedure; however, the Boomerang device is used in almost all of our patients undergoing a neuro imaging or treatment procedure. The neuroradiologist will determine which device if any is best for you based on the size of your artery, your medical condition etc. We will only collect data about you and your procedure if the Boomerang device is used.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that has a percutaneous Boomerang closure device placed after having a neuro-intervention

Exclusion Criteria:

* Patients that do not have this medical device used post procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having a neurointerventional procedure, such as a cerebral angiography
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States